CLINICAL TRIAL: NCT02929914
Title: Effect of Antimicrobial Photodynamic Therapy on Deep Caries in Permanent Tooth: A Pilot Randomized Controlled Trial
Brief Title: Effect of aPDT on Deep Caries in Permanent Tooth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xiaojing Huang, DDS, PhD, Professor，Vice Dean，School and Hospital of Stomatology Fujian Medical University, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDT20160602
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Dental Caries
Keywords: Carious dentin; Photodynamic Therapy
MeSH Terms: conditions — Dental Caries | interventions — Anesthesia, Local; Sodium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Experimental): Local anesthesia, rubber dam isolation, remove caries incompletely, microbiological sample with otoscope curette, dentin washed with sodium 0.9% saline, sampling again. Indirect pulp treatment with calcium hydroxide(CH). Restoration with resin(Z350,3M). Follow up at 6, 12 and 24 months.
  Interventions: Procedure: Local anesthesia and rubber dam isolation; Procedure: Incomplete caries removal and microbiological samples collection; Procedure: Dentin washed with sodium 0.9% saline; Procedure: Microbiological samples collection and Indirect pulp treatment
- PDT+CH (Experimental): Local anesthesia, rubber dam isolation, remove caries incompletely, microbiological sample with otoscope curette, disinfect the remaining dentin with antimicrobial photodynamic therapy (DENFOTEX PADplus), sampling again. Indirect pulp treatment with calcium hydroxide(CH). Restoration with resin(Z350,3M). Follow up at 6, 12 and 24 months.
  Interventions: Procedure: Local anesthesia and rubber dam isolation; Procedure: Incomplete caries removal and microbiological samples collection; Procedure: Antimicrobial Photodynamic Therapy; Procedure: Microbiological samples collection and Indirect pulp treatment

INTERVENTIONS:
Procedure: Local anesthesia and rubber dam isolation — Local anesthesia was performed. Tooth was isolated using a rubber dam isolation in order to collect the dentin samples.
Procedure: Incomplete caries removal and microbiological samples collection — Partial carious tissue was removed with conventional dentinal curette and collection of dentin with a spoon (1#) was performed.
Procedure: Dentin washed with sodium 0.9% saline — The remaining dentin was dipped in sodium 0.9% saline for 2min.
  Arms: Control
Procedure: Antimicrobial Photodynamic Therapy — The remaining dentin was disinfected with aPDT for 2 min.
  Arms: PDT+CH
Procedure: Microbiological samples collection and Indirect pulp treatment — A new dentin collection was performed after this treatment at another site of the cavity. Then teeth were conventionally restored using the following materials: calcium hydroxide lining material and resin (Z350,3M).

SUMMARY:
The aim of this study is to assess the clinical effect of aPDT on deep caries in permanent teeth. Half of the deep caries will receive aPDT disinfect in restorative treatment procedure, while the other half will receive sodium 0.9% saline in restorative treatment procedure.

DETAILED DESCRIPTION:
The aim of the proposed study is to assess the clinical effect of antimicrobial photodynamic therapy (aPDT) using LED on dentin with deep caries in permanent teeth. Permanent teeth with deep carious lesions on the occlusal surface indicated for restorative treatment will be randomly allocated to two groups: Group 1 -Control after incomplete caries removal, washed with sodium 0.9% saline; Group 2 - PDT + CH after incomplete caries removal, disinfect the residual dentin with PDT(LED + O-Toluidine Blue). Dentin samples will be collected before and after disinfect for microbiological analysis. Then the teeth will be capped with CH and restored using resin with clinical and radiographic follow up at 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Good general health, without syndromes or chronic systemic diseases
* Permanent tooth with deep carious lesion (2/3 of dentin) without pain symptomatology and compatible with reversible pulpits

Exclusion Criteria:

* Refused to sign the informed consent document
* Allergic to photosensitizer
* Unlikely to be able to comply with the study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of bacteria by colony counting | 2 days after dentin collection
  Quantification of total bacteria

SECONDARY OUTCOMES:
Tooth Pain | 1 day and 6, 12, 24 months
  Patients reported the presence or absence of tooth pain
Restoration Quality | 1 day and 6, 12, 24 months
  The quality of restoration was evaluated through the absence of radiographic radiolucent area

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Huang, PhD, Study Chair — School and Hospital of stomatology, Fujian Medical University
Locations (1):
- School and Hospital of Stomatology, Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No